CLINICAL TRIAL: NCT07383493
Title: Evaluation of Treatments for Acute Viral Rhinitis, Rhinosinusitis, and Rhinopharyngitis
Brief Title: RhinAV_Evaluation of Treatments for Acute Viral Rhinitis, Rhinosinusitis, and Rhinopharyngitis
Acronym: RhinAV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RBHP 2025 PICKERING 4
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Rhinitis Acute; Rhinitis Viral; Rhinosinusitis Acute; Rhinopharyngitis; Rhinitis; Rhinosinusitis
MeSH Terms: conditions — Common Cold; Nasopharyngitis; Rhinitis; Rhinosinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PIR (Experimental): Patients included in the "PIR" arm will receive the medical device of the same name.
  Interventions: Device: PIR
- NS (Experimental): Patients included in the "NS" arm will receive the medical device of the same name.
  Interventions: Device: NS
- NHE (Experimental): Patients included in the "NHE" arm will receive the medical device of the same name.
  Interventions: Device: NHE
- NHG (Experimental): Patients included in the "NHG" arm will receive the medical device of the same name.
  Interventions: Device: NHG

INTERVENTIONS:
Device: PIR — Patients included in the "PIR" arm will receive the medical device of the same name.
  Arms: PIR
Device: NS — Patients included in the "NS" arm will receive the medical device of the same name.
  Arms: NS
Device: NHE — Patients included in the "NHE" arm will receive the medical device of the same name.
  Arms: NHE
Device: NHG — Patients included in the "NHG" arm will receive the medical device of the same name.
  Arms: NHG

SUMMARY:
The objective of this study is to conduct post-marketing clinical follow-up of four products: NS, NHE, NHG, and PIR. This follow-up will consist of collecting clinical data in real-life conditions to confirm the tolerance, safety, and efficacy of medical devices used in the treatment of acute viral rhinitis, rhinosinusitis, and rhinopharyngitis, while also assessing the benefit/risk ratio of the products.

ELIGIBILITY:
Inclusion Criteria:

* Acute viral rhinitis or acute rhinosinusitis or viral rhinopharyngitis (sneezing, rhinorrhea, nasal obstruction, cough secondary to posterior rhinorrhea, sore throat) that began less than 72 hours prior to the inclusion visit, in the investigator's judgment,
* Effective contraception for female patients of childbearing age.
* Cooperation and sufficient understanding to comply with the requirements of the trial.
* Acceptance of registration in the SI-RIPH VRB file.
* Having received informed information and agreeing to give written consent.
* Affiliated with the French Social Security system.

Exclusion Criteria:

* Hypersensitivity/history of allergy to any of the product's components,
* Complicated rhinitis, rhinosinusitis, or rhinopharyngitis (acute bacterial sinusitis, acute otitis media, acute bronchitis, or pneumonia) or severe cough that is poorly tolerated,
* Chronic rhinosinusitis,
* Allergic rhinosinusitis,
* Other ongoing treatments for acute rhinitis (local treatment, antitussives, antibiotics, antiretrovirals, corticosteroids, etc.),
* Positive antigen test for influenza A/B or COVID-19 and infection requiring etiological treatment according to the recommendations,
* Bacterial rhinopharyngitis with positive TROD test
* Comorbidities or health conditions deemed incompatible with the trial by the investigator,
* Recent ENT surgery (<6 months),
* ENT pathology such as nasal septum deviation or other causes of nasal obstruction,
* Pulmonary pathology (COPD, asthma, etc.),
* Immunosuppression (as reported by the patient),
* Pregnant or breastfeeding women,
* Currently participating in another clinical trial, or in the exclusion period, or having received total compensation of more than €6,000 in the 12 months prior to the start of the trial,
* Benefiting from legal protection measures (guardianship, trusteeship, deprivation of liberty, judicial protection).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Tolerance | From visit 1 (day 1) to visit 2 (day 15)
  Collection of adverse events (AEs) during the period of use of PIR, NS, NHE, and NHG products in an electronic daily recording book.

SECONDARY OUTCOMES:
Efficiency | From visit 1 (day 1) to the last day of use of the study product (day 14)
  Clinical improvement (yes/no) defined as a decrease of at least 30% in the "total score for symptoms of rhinitis, rhinosinusitis, and rhinopharyngitis" (STS3R) between baseline and the average of the scores measured during the last 3 days of use of the study product (days 12, 13, and 14).
Quality of life impact | From visite 1 (day 1) to visit 2 (day 15)
  Change in quality of life measured by four questions before (Day 1) and after (Day 15) use of the study products concerning sleep, daily activities, fatigue, and irritability. Each response will be rated between 0 (not impacted) and 10 (highly impacted) on a visual analog scale.
Device defect | From visit 1 (day 1) to visit 2 (day 15)
  Device defect assessed by recording any defect in terms of identity, quality, durability, reliability, safety, or performance, malfunction, or user error, or any defect in the information provided by the manufacturer in the electronic record book.

CONTACTS AND LOCATIONS:
Overall Officials: Lise Laclautre, Study Chair — University Hospital, Clermont-Ferrand
Locations (1):
- Plateforme d'investigation clinique/Centre d'Investigation Clinique, Inserm CIC 1405, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Undecided